CLINICAL TRIAL: NCT01925625
Title: Detection in Blood of Autoantibodies to Tumour Antigens as a Case-finding Method in Lung Cancer Using the EarlyCDT-Lung Test
Brief Title: Early Cancer Detection Test - Lung Cancer Scotland
Acronym: ECLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stuart Schembri (Other)
Responsible Party: Sponsor-Investigator, Stuart Schembri, Consultant, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2013ON07
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): participants monitored for 10 years for lung cancer incidence.
- Early CDT Lung Test (Active Comparator): Early CDT lung blood test
  Interventions: Biological: Early CDT Lung blood test

INTERVENTIONS:
Biological: Early CDT Lung blood test — The EarlyCDT-Lung Test is an early detection test designed to assist in lung cancer risk assessment and detection in the earliest stages of the disease.
  Other Names: EarlyCDT-Lung test
  Arms: Early CDT Lung Test

SUMMARY:
HYPOTHESIS In a high risk population the EarlyCDT-Lung test reduces the incidence of late stage tumours;3 / 4 / Unclassified (U) at diagnosis compared to normal clinical practice.

DETAILED DESCRIPTION:
AIMS To assess the effectiveness of EarlyCDT-Lung test in increasing early stage lung cancer detection, thereby reducing the rate of late stage (3 / 4 / U) presentation, compared to normal clinical practice; to assess the cost-effectiveness of EarlyCDT-Lung test compared to normal clinical practice; to assess the effectiveness of EarlyCDT-Lung test in reducing adverse outcomes including potential psychological and behavioural consequences.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study
2. Male or female aged 50 years to 75 years
3. Current or Ex-smoker with at least 20 year pack history
4. or Less than 20 year pack history but with family history of lung cancer in a 1st degree relative (mother, father, sister, brother, child)
5. ECOG Status: 0, 1 and 2 (Eastern Co-operative Oncology Group) Grade ECOG 0 Fully active, able to carry on all pre-disease performance without restriction 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work 2 Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
6. Geographical postal sectors of:

NHS Geographical Area Eligible Postcodes Tayside DD1 - DD11, PH1-PH3 , PH6-PH8, PH10, PH11, PH13, PH15 & PH16 Greater Glasgow & Clyde G1-G5, G11 -G15, G20-G22, G31-34, G40 -G46, G51- G53, G60-G62 &G64, G66 & G69, G72 & G73, G76-G78, G81-G83 PA1-PA8 (except PA6), PA11-PA16 & PA19

Exclusion Criteria:

1. History of any cancer other than non-melanomatous skin cancer, cervical cancer in situ.
2. Symptoms suggestive of lung cancer within past 6 months (haemoptysis, unintentional weight loss (at least 5% in preceding 6 months).
3. Patients for whom the GP considers invitation to the study would cause undue distress.
4. Patients with other terminal disease.
5. Patients on prolonged / continuous use (> 3months) of cytotoxic/ immuno-suppressant drugs eg: Cyclophosphamide. Monotherapy using glucocorticoids/ steroids eg prednisolone is NOT an exclusion criteria.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12210 (Actual)
Dates: Start 2013-08; Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
to assess the effectiveness of EarlyCDT-Lung test in reducing the incidence of patients with late-stage lung cancer at diagnosis, compared with standard clinical practice; | 24 months
  difference at 24 months after randomisation, between the number of patients with stage 3, 4 or unclassified lung cancer at diagnosis in the intervention arm, and those in the control arm;

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sullivan, MbChB, Principal Investigator — University of Dundee
Locations (3):
- United Kingdom (3):
  - NHS Tayside, Dundee, Tayside
  - NHS Greater Glasgow & Clyde, Glasgow
  - NHS Lanarkshire, Wishaw

IPD SHARING:
Plan to Share IPD: Undecided
paticipant activity nearing closure

REFERENCES:
- [Derived] Romeikat NL, Sullivan F, Daly F, Kong W. The Importance of Comorbidities at Baseline and 5-Year Follow-Up in a Lung Cancer Biomarker Screening Trial. J Clin Med. 2025 Mar 20;14(6):2116. doi: 10.3390/jcm14062116. PMID 40142924
- [Derived] Madurasinghe VW, Bower P, Eldridge S, Collier D, Graffy J, Treweek S, Knapp P, Parker A, Rick J, Salisbury C, Man MS, Torgerson D, Sheridan R, Sullivan F, Cockayne S, Dack C. Can we achieve better recruitment by providing better information? Meta-analysis of 'studies within a trial' (SWATs) of optimised participant information sheets. BMC Med. 2021 Sep 23;19(1):218. doi: 10.1186/s12916-021-02086-2. PMID 34551765
- [Derived] Sullivan FM, Mair FS, Anderson W, Armory P, Briggs A, Chew C, Dorward A, Haughney J, Hogarth F, Kendrick D, Littleford R, McConnachie A, McCowan C, McMeekin N, Patel M, Rauchhaus P, Ritchie L, Robertson C, Robertson J, Robles-Zurita J, Sarvesvaran J, Sewell H, Sproule M, Taylor T, Tello A, Treweek S, Vedhara K, Schembri S; Early Diagnosis of Lung Cancer Scotland (ECLS) Team. Earlier diagnosis of lung cancer in a randomised trial of an autoantibody blood test followed by imaging. Eur Respir J. 2021 Jan 14;57(1):2000670. doi: 10.1183/13993003.00670-2020. Print 2021 Jan. PMID 32732334
- [Derived] Parker A, Knapp P, Treweek S, Madhurasinghe V, Littleford R, Gallant S, Sullivan F, Schembri S, Rick J, Graffy J, Collier DJ, Eldridge S, Kennedy A, Bower P. The effect of optimised patient information materials on recruitment in a lung cancer screening trial: an embedded randomised recruitment trial. Trials. 2018 Sep 18;19(1):503. doi: 10.1186/s13063-018-2896-9. PMID 30227890
- [Derived] Sullivan FM, Farmer E, Mair FS, Treweek S, Kendrick D, Jackson C, Robertson C, Briggs A, McCowan C, Bedford L, Young B, Vedhara K, Gallant S, Littleford R, Robertson J, Sewell H, Dorward A, Sarvesvaran J, Schembri S. Detection in blood of autoantibodies to tumour antigens as a case-finding method in lung cancer using the EarlyCDT(R)-Lung Test (ECLS): study protocol for a randomized controlled trial. BMC Cancer. 2017 Mar 11;17(1):187. doi: 10.1186/s12885-017-3175-y. PMID 28284200
- See also: Study website — http://www.eclsstudy.org